CLINICAL TRIAL: NCT05831423
Title: The Role of Licensing in Early Care and Education (TRLECE): Survey of State Front-Line Licensing Staff
Brief Title: The Role of Licensing in Early Care and Education: Front-Line Licensing Staff
Acronym: TRLECE: FLLS
Status: Completed | Type: Observational
Sponsor: Child Trends (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); ICF International, Inc. (Unknown)
Responsible Party: Principal Investigator, Kelly Maxwell, Senior Researcj Scholar, Early Childhood Research, Child Trends
Other Study IDs: 17187002; 233201500034I-75P00119F37007 (Other Grant/Funding Number: OPRE, ACF, US Dept. Health and Human Services (HHSP))
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Licensing Staff Perceptions of the Licensing System
Keywords: Child care and early education; Child care licensing; Early care and education programs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Child Trends, funded by the Office of Planning, Research, and Evaluation, Administration for Children and Families (ACF) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for The Role of Licensing in Early Care and Education (TRLECE): Front-Line Licensing Staff project. The goal of this information collection is to deepen the field's understanding of child care and early education licensing systems, which play a critical role in supporting positive outcomes for providers, families, and children. The investigators will conduct one round of survey data collection with front-line child care licensing staff in all states.

DETAILED DESCRIPTION:
This study aims to advance understanding of the landscape of child care and early education licensing systems. State/territory child care and early education licensing agencies establish and monitor regulations that child care programs serving young children must meet to operate legally. These regulations and monitoring practices play a large role in the operations of child care programs but have received relatively little research attention. The field has limited information about features of state/territory licensing units; and no information directly from front-line licensing staff about their characteristics, experiences, training, and perceptions of licensing. Ultimately, TRLECE: Front-Line Licensing Staff findings can inform licensing policies, practices, and supports in the child care and early education field; guidance and technical assistance to state leaders; and future research.

The investigators will conduct a survey of front-line child care licensing staff, who are the individuals who routinely conduct inspections of licensed child care programs, for this descriptive study. The survey is designed to collect information about front-line staff members' roles, day-to-day responsibilities, demographic characteristics, career paths, professional development experiences, relationships with colleagues and providers, and burnout/work satisfaction, role in supporting quality and quality improvement, and perceptions of strengths and challenges of the licensing system. The investigators intend to invite all front-line staff from all 50 states and DC to participate (n=~3,000).

ELIGIBILITY:
Inclusion Criteria:

* All front-line child care licensing staff in all U.S. states and DC

Exclusion Criteria:

* Individuals who are not front-line child care licensing staff in U.S. states and DC

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Front-line child care licensing staff
Sampling Method: Non-Probability Sample
Enrollment: 1159 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Front-line child care licensing staff survey | one time
  Survey developed by the study team to gather child care front-line licensing staff's demographic characteristics, background and experiences, job duties, perceptions of their role, burnout, relationships with providers, and ideas for improving licensing

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Maxwell, PhD, Principal Investigator — Child Trends
Locations (1):
- Child Trends Headquarters, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD collected in the survey will be shared with the Child & Family Data Archive (CFData).
Time Frame: The team anticipates submitting IPD and supporting information to Child and Family Data Archive (CFData) roughly 6 months after the end of data collection. Data will be available after being reviewed by CFData. No end date on the availability of the data.
Access Criteria: Most data from the front-line staff survey will be archived as public-use data with CFData and accessible on their website. Some data will be available as restricted-use only, following guidelines from CFData. Data will be shared with researchers for analyses related to child care licensing practices and experiences of front-line staff.